CLINICAL TRIAL: NCT03452891
Title: Effect of Locally-Applied Simvastatin on Clinical Attachment Level and Alveolar Bone in Periodontal Maintenance Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0217-18-FB
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Results first posted 2023-02-09 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Methylcellulose; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Simvastatin Methylcellulose (Experimental): simvastatin in methylcellulose gel
  Interventions: Drug: Simvastatin-Methylcellulose
- Methylcellulose Gel (Placebo Comparator): Methylcellulose gel
  Interventions: Other: Methylcellulose

INTERVENTIONS:
Other: Methylcellulose — Methylcellulose gel will be placed in a deep (6-9 mm) periodontal pocket.
  Arms: Methylcellulose Gel
Drug: Simvastatin-Methylcellulose — Simvastatin-Methylcellulose gel will be placed in a deep (6-9 mm) periodontal pocket.
  Other Names: Simvastatin
  Arms: Simvastatin Methylcellulose

SUMMARY:
The purpose of this study is to determine of local application of commericially-available, FDA-approved preparation of simvastatin is effective in increasing clinical attachment levels (primary outcome), as well as alveolar bone (secondary outcome) compared to standard mechanical therapy in patients on periodontal maintenance therapy (PMT). Subjects undergoing PMT at the UNMC College of Dentistry clinics will be recruited to participate in the randomized one-year clinical trial based on the following eligibility criteria: 1) diagnosis of chronic advanced periodontitis (generalized or localized), 2) participating in regular PMT visits (3-6) month intervals), 3) no systemic diseases or medication which significantly impact periodontal inflammation or bone turnover (e.g. steroids, bisphosphonates, > 325 mg aspirin/day and in good general health, 4) one experimental quadrant of the mouth with an inflamed 6-9 mm interproximal posterior periodontal pocket with history of bleeding on probing (BOP), 5) willingness to sign consent form. Subjects will be divided into two groups for additional therapy in a 6-9 mm interproximal periodontal pocket at baseline: 1) local anesthesia and mini-flap reflection with subgingival mechanical debridement plus application of the simvastatin-methylcellulose gel or 2) local anesthesia and mini-flap reflection with subgingival mechanical debridement plus application of methylcellulose gel alone. Samples/measurement will be obtained at the designated experimental site at baseline, 2 weeks, 6 and 12 months during PMT: 1) digital radiographs (baseline and 12 months only; bone height measurements), 2) presence of explorer-detectable supragingival plaque, 3) 30-second gingival crevicular fluid (GCF) sample (markers of inflammation, bone turnover), 4) recession from the cemento-enamel junction, 5) probing pocket depth and bleeding on probing (BOP). Following the 12-month visit, the research-specific intervention and measurements in the experiment quadrant will be removed from routine PMT.

DETAILED DESCRIPTION:
Dental records of patients attending routine periodontal maintenance therapy visits at the UNMC College of Dentistry clinics are reviewed as part of the direct supervision by faculty, including investigators involved int his study. Assessment includes review of medical and dental histories and previous oral hygiene and periodontal charting. Subjects who appear to qualify (40-85 years old, diagnosis of advanced chronic adult periodontitis, one quadrant with at least 3 posterior teeth and one 6-9 mm periodontal pocket, no systemic diseases or medications which significantly impact periodontal inflammation and bone turnover) will be informed of the study, given an opportunity to ask questions, and given an informed consent form to take home. Once signed consent is obtained, subjects will be randomized to one of the two groups: 1) SRP + SIM or 2) SRP + methylcellulose.

At the baseline visit, all women subjects will be given a urine pregnancy test. Once the pregnancy test is determined to be negative, the following sequence of procedures will be performed by the faculty investigator (AK, RR, RH): 1) assignment of the experimental site (6-9 mm pocket with previous bleeding on probing); 2) remove supraginigval plaque from the experimental tooth with explorer [record positive sites]; 3) insert paper strip into facial and lingual of experimental site sulcus for 30 seconds for gingival crevicular fluid (GCF) sample, remove and place into sterile vial, and freeze at -80º C for testing inflammation markers; 4) measure recession on experimental teeth and adjacent interproximal tooth at mesial-facial, mid-facial, distal-facial, mesial-lingual, mid-lingual and distal lingual with UNC 15 probe; 5) measure probing pocket depths at same surfaces as recession; 6) record sites that bleed within 30 seconds. After the faculty investigator (primary or secondary investigator) leaves, the participating personnel (LK) will; 7) take a baseline radiograph, administer local anesthesia to the experimental site via local injection, 9) surgical mini-flap reflection localized to the experimental site (papilla reflection), 10) remove most of the remaining interproximal soft tissue to allow access to the root and measure markers of inflammation, 11) scaling/root planing of site to remove supra- and subgingival bacterial plaque and calculus; 12) placement of SIM-methylcellulose gel, 13) repositioning of papilla to initial location and placement of intra-oral cyanoacrylate; 14) finish full-mouth measurement of probing depths and bleeding on probing; 15) perform full-mouth scaling to remove supra- and subgingival bacterial plaque and calculus; 16) review oral hygiene instructions.

It is possible that steps 14, 15 and 16 could be completed prior to steps 1-13 on all teeth except experimental and adjacent teeth due to availability of faculty investigators at the time of the PMT appointment.

It is also possible that steps 1-13 could be completed at a separate appointment.

Subjects will return for postoperative visit in two weeks. Subjects will return for subsequent PMT visits after 3, 6, 9 and 12 months. Steps 14-16 will be completed at each visit as part of routine PMT. At 6 and 12 months, steps 2-6 will also be completed. At 12 months, a radiograph will also be taken.

Dental record data that will be recorded at each visit includes probing depths (PD), recession, bleeding on probing (BOP) and presence of plaque (+/-) at test site and adjacent interproximal sites.

The expected amount of time for the baseline visit in 90-120 minutes. The expected amount of time for subsequent visits in 60-90 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. age 40-85 years,
2. diagnosis of chronic advanced adult periodontitis,
3. one quadrant with at least one 6-9 mm interproximal pocket,
4. overall good systemic health,
5. willingness to sign consent form.

Exclusion Criteria:

1. systemic diseases which significantly impact periodontal inflammation and bone turnover (e.g. rheumatoid arthritis),
2. taking drugs which significantly impact periodontal inflammation and bone turnover (e.g. chronic use of steroids or non-steroidal anti-inflammatory drug (>325 mg/d), estrogens, bisphosphonates, calcitonin, methotrexate),
3. surgical periodontal therapy within the past year,
4. pregnant or breast-feeding females.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Killeen, DDS, MS, Principal Investigator — University of Nebraska Medical Center College of Dentistry
Locations (1):
- University of Nebraska, College of Dentistry, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SIM-MCL: Simvastatin-Methylcellulose: Simvastatin-Methylcellulose gel will be placed in a deep (6-9 mm) periodontal pocket.
Period: Overall Study
Arm/Group | SIM-MCL | Methylcellulose Gel
Started | 25 (25 subjects) | 25
Subjects Enrolled | 25 | 25
Subjects Completing Study | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Fifty periodontal maintenance subjects with chronic inflammation participated in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | SIM-MCL | Methylcellulose Gel | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 20 | 37
  >=65 years | 8 | 5 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 7 | 5 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Attachment Level (CAL)
Description: The change in CAL will be measured and calculated by measuring recession and subtracting the periodontal probing depth.
Time Frame: The CAL will be measured at 12-months.
Measure: Mean (Standard Error); unit: millimeters
Arm/Group | SIM-MCL | Methylcellulose Gel
Number analyzed (Participants) | 25 | 25
millimeters | 7.0 (0.1) | 6.9 (0.2)

ADVERSE EVENTS:
Time Frame: 1 year, 9 months
Description: All-cause mortality was 0/50, or 0/25 for each arm of study. Thus risk of all-cause mortality was 0.
  Serious adverse events was 0/50, or 0/25 for each arm of study, thus risk of serious adverse events was 0.
  Other adverse events was 0/50, or 0/25 for each arm of study. Thus risk of Other adverse events was 0.
Arm/Group | SIM-MCL | Methylcellulose Gel
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT03452891/Prot_SAP_002.pdf